CLINICAL TRIAL: NCT02407899
Title: A Randomized Controlled, Open-label, Multi-center Study With 104-week Saxagliptin or (and) Vitamin D3 Assessing Protective Effects on Beta Cell Function in Latent Autoimmune Diabetes in Adults (LADA) Treated With Metformin (and Insulin)
Brief Title: Protective Effects of Saxagliptin (And Vitamin D3) on β Cell Function in Adult-onset Latent Autoimmune Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Beijing Hospital (Other Government); The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, Director, Department of Endocrinology, Institute of Metabolism and Endocrinology, National Clinical Research Center for Metabolic Diseases, Second Xiangya Hospital, Central South University, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCRCMD LADA SAX 2015
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: LADA; saxagliptin; vitamin D3; C-Peptide
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — saxagliptin; Dipeptidyl Peptidase 4; Cholecalciferol; Insulin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- Metformin (and insulin) + saxagliptin (Experimental): Patients who have diagnosed LADA are assigned to receive Saxagliptin tablets 5mg/d and Metformin 1.5g/d (and insulin at individual dose) for 104-week.
  Interventions: Drug: Saxagliptin; Drug: Insulin; Drug: Metformin
- Metformin(insulin)+saxagliptin +vitamin D3 (Experimental): Patients who have diagnosed LADA are assigned to receive Saxagliptin tablets 5 mg/d, vitamin D drop 2000IU/d, Metformin 1.5g/d (and insulin at individual dose) for 104-week.
  Interventions: Drug: Saxagliptin; Drug: Vitamin D3; Drug: Insulin; Drug: Metformin
- Metformin (and insulin) (Active Comparator): Patients who have diagnosed LADA are assigned to receive Metformin 1.5g/d(and insulin at individual dose) for 104-week.
  Interventions: Drug: Insulin; Drug: Metformin

INTERVENTIONS:
Drug: Saxagliptin — Take saxagliptin tablet 5mg p.o. qd. for 104 weeks after randomization.
  Other Names: Onglyza; Dipeptidyl peptidase 4 (DPP-4) inhibitor
  Arms: Metformin (and insulin) + saxagliptin; Metformin(insulin)+saxagliptin +vitamin D3
Drug: Vitamin D3 — Take vitamin D drops 2000 IU p.o. qd. for 104 weeks after randomization.
  Other Names: Cholecalciferol
  Arms: Metformin(insulin)+saxagliptin +vitamin D3
Drug: Insulin — For optimal control of patients' glucose, researchers can initiate insulin therapy at any time in this trial, choose any brands of insulin after discussion with the patient.
  Other Names: Recombinant Human Insulin, Insulin analogue.
Drug: Metformin — Take Metformin tablet 1.5g p.o. per day for 104 weeks (adjust the dose between 1-1.7g per day according to subject's specific situation) before or after randomization.
  Other Names: Metformin Hydrochloride tablet

SUMMARY:
The main purpose of this study is to evaluate whether saxagliptin or (and vitamin D3) with metformin (and insulin) therapy can better protect islet β cell function than metformin(and insulin) .

DETAILED DESCRIPTION:
LADA is actually a form of type 1 diabetes, which is caused by autoimmune damage of islet β cells and triggered by environmental factors based on genetic susceptibility. LADA shows some characteristics of type 2 diabetes at its onset, which develops slowly and latent, and easily be misdiagnosed as type 2 diabetes due to slowly β cell function deterioration. This is a multi-center, open- label, 1:1:1 randomized controlled trial to investigate the protective effects of saxagliptin and vitamin D3 in LADA patients. The study comprises the 0-6weeks of screening period and the 104-week intervention period. After obtaining the informed consent，the screening will find out the eligible patients according to the inclusion/exclusion criteria, then the patients will be randomized to the 104-week intervention period. Subjects will be randomized into one of the three groups(arms) through central dynamic randomization: metformin (and insulin), metformin(and insulin) +saxagliptin, metformin(and insulin) +saxagliptin+vitamin D3. Our previous randomized- controlled pilot study showed that dipeptidyl peptidase 4 (DPP-4) inhibitors could significantly improve islet β-cell function in patients with LADA. The main purpose of this study: To evaluate whether saxagliptin (and vitamin D3) with metformin (and insulin) therapy can better protect islet β cell function than metformin (and insulin).

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study with informed consent;
2. The LADA patients to be included in this study are defined as:

(1) Meet the 1999 WHO Diagnostic Criteria for Diabetes Mellitus; (2) Age at diagnosis of DM ≧ 18 years old; (3) Glutamic acid decarboxylase antibody (GADA) positive; (4) Serum fasting C-peptide ≥ 100 pmol/L or 2-hour postprandial C-peptide≥ 200 pmol/L; 3. Age between 18-70 years old; 4. Diabetes duration <4 year; 5. Outpatient or inpatient.

Exclusion Criteria:

1. Pregnancy, breastfeeding or planned pregnancy within two years;
2. Gestational diabetes mellitus or other specific types of diabetes;
3. Allergic to saxagliptin, vitamin D3 and their excipient;
4. Treatment with any anti-diabetic medication other than insulin in the last 8 weeks prior to randomization;
5. Use of systemic corticosteroids therapy (oral, intravenous) continuously for more than 7 days over the past 6 months;
6. Treatment with cytochrome P450 3A4/5 (CYP450 3A4/5) inhibitor;
7. Alanine aminotransferase (ALT) or aspartate transaminase(AST) more than 3 times of the normal upper limit, total bilirubin (TBIL) more than 2 times of the normal upper limit;
8. Creatinine levels ≧ 1.5 mg/dL(132μmol/L) for males and ≧ 1.4 mg/dL (123μmol/L) for females or creatinine clearance ≦ 50 mL/min;
9. History of malignant tumors;
10. History of mental disorders;
11. History of alcohol abuse or illegal drug abuse;
12. Serious systemic disease which the investigators think would not be suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-03; Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Absolute changes from baseline in Fasting C-peptide levels at week 104. | From baseline to 104 week
  1. To evaluate the efficacy of saxagliptin plus metformin (and insulin) on beta cell function in LADA patients compared with metformin (and insulin) treatment. By measure absolute changes from baseline in Fasting C-peptide levels at week 104.
  2. To evaluate the efficacy of saxagliptin (add on vitamin D) plus metformin (and insulin) on beta cell function in LADA patients compared with metformin (and insulin) treatment.By measure absolute changes from baseline in Fasting C-peptide levels at week 104.

SECONDARY OUTCOMES:
Absolute changes from baseline in fasting C-peptide levels and at week 26, 52 and 78. | From baseline to 26, 52, 78 week
  To evaluate the efficacy of saxagliptin (add on vitamin D) plus metformin (and insulin) on indicators of beta cell function compared with LADA patients treated with metformin (and insulin). By measure absolute changes from baseline in fasting C-peptide levels and at week 26, 52 and 78.
Absolute changes from baseline in C peptide at 60-min and 120-min (AUC) during a mixed-meal tolerance test and at week 26, 52, 78 and 104. | From baseline to 26, 52, 78, 104 week
  To evaluate the efficacy of saxagliptin (add on vitamin D) plus metformin (and insulin) on indicators of beta cell function compared with LADA patients treated with metformin (and insulin). By measure absolute changes from baseline in C peptide at 60-min and 120-min (AUC) during a mixed-meal tolerance test and at week 26, 52, 78 and 104.
The proportion of subjects with increased (decreased, unchanged) fasting or post-stimulus C peptide level compared with baseline after 104 weeks of treatment. | From baseline to 104 week
  To evaluate the efficacy of saxagliptin (add on vitamin D) plus metformin (and insulin) on indicators of beta cell function compared with LADA patients treated with metformin (and insulin). By measure the proportion of subjects with increased (decreased, unchanged) fasting or post-stimulus C peptide level compared with baseline after 104 weeks of treatment.
The increased percentage of C peptide pre-and post mixed-meal tolerance test (Delta C peptide) after 104 weeks of treatment. | From baseline to 104 week
  To evaluate the efficacy of saxagliptin (add on vitamin D) plus metformin (and insulin) on indicators of beta cell function compared with LADA patients treated with metformin (and insulin). By measure the increased percentage of C peptide pre-and post mixed-meal tolerance test (Delta C peptide) after 104 weeks of treatment
Changes of HbA1c levels from baseline and at week 26, 52, 78 and 104. | 26, 52, 78, 104 week
  To evaluate the efficacy of saxagliptin (add on vitamin D) plus metformin (and insulin) on glycemic control compared with LADA patients treated with metformin (and insulin). By measure Changes of HbA1c levels from baseline and at week 26, 52, 78 and 104.
The proportion of subjects responding to glucose therapy (i.e. HbA1c<7%) after 104 weeks of treatment. | 104 week
  To evaluate the efficacy of saxagliptin (add on vitamin D) plus metformin (and insulin) on glycemic control compared with LADA patients treated with metformin (and insulin). By measure the proportion of subjects responding to glucose therapy (i.e. HbA1c<7%) after 104 weeks of treatment.
Changes of average daily insulin dose (U/kg/d) from baseline and at week 26, 52, 78 and 104 | From baseline to 26, 52, 78, 104 week
  To evaluate the efficacy of saxagliptin (add on vitamin D) plus metformin (and insulin) on glycemic control /insulin-sparing compared with LADA patients treated with metformin (and insulin). By measure Changes of average daily insulin dose (U/kg/d) from baseline and at week 26, 52, 78 and 104.
Changes of GADA titers from baseline and at week 52 and 104. | From baseline to 52, 104 week
  To evaluate the efficacy of saxagliptin (add on vitamin D) plus metformin (and insulin) on glycemic control /insulin-sparing/changes of autoantibody titer compared with LADA patients treated with metformin (and insulin). By measure changes of GADA titers from baseline and at week 52 and 104.
Absolute changes of body weight and BMI level from baseline and at week 26, 52, 78 and 104. | From baseline to 26, 52, 78, 104 week
  To evaluate the efficacy of saxagliptin (add on vitamin D) plus metformin (and insulin) on body weight/BMI level compared with LADA patients treated with metformin (and insulin). By measure Changes of BMI from baseline and at week 26, 52, 78 and 104.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguang Zhou, MD/PhD, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (39):
- China (39):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Hospital of the Ministry of Health, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Quanzhou First Hospital, Fujian, Quanzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fujian, Fuzhou
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - Tangshan Gongren Hospital063000, Tangshan, Hebei
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First People's Hospital of Changde, Changde, Hunan
  - Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Affiliated Hospital of South China University, Hengyang, Hunan
  - The Second Hospital University of South China, Hengyang, Hunan
  - The First People's Hospital of Huaihua, Huaihua, Hunan
  - The First People's Hospital of Yueyang, Yueyang, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Third Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Jilin Province People's Hospital, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality
  - Heping Hospital of Changzhi Medical College, Changzhi, Shanxi
  - Affiliated Heji Hospital of Changzhi Medical College, Changzhi, Shanxi
  - The First Affiliated Hospital of The Fourth Military Medical University, Xi’an, Shanxi
  - First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Yan X, Li X, Liu B, Huang J, Xiang Y, Hu Y, Tang X, Zhang Z, Huang G, Xie Z, Zhou H, Liu Z, Wang X, Leslie RD, Zhou Z. Combination therapy with saxagliptin and vitamin D for the preservation of beta-cell function in adult-onset type 1 diabetes: a multi-center, randomized, controlled trial. Signal Transduct Target Ther. 2023 Apr 20;8(1):158. doi: 10.1038/s41392-023-01369-9. PMID 37076476